CLINICAL TRIAL: NCT03025581
Title: Does Nipple Stimulation Shorten Time to Vaginal Birth in Women With Term PROM? (NIPROM Study)
Brief Title: Does Nipple Stimulation Shorten Time to Vaginal Birth in Women With Term PROM?
Acronym: NIPROM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 0091-HYMC
Record Dates: First submitted 2017-01-06; First posted 2017-01-19 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Premature Rupture of Fetal Membranes
MeSH Terms: conditions — Fetal Membranes, Premature Rupture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Active Comparator): Nipple stimulation.
  Interventions: Other: Nipple stimulation
- Control group (No Intervention): No intervention (expectant management only).

INTERVENTIONS:
Other: Nipple stimulation — For the intervention group participants will be instructed to gently massage alternate breasts, especially around the nipples for 15 minutes every 6 hours until the appearance of regular contractions but not more than 24 hours. Moist cloth or lubricating or moisturizing cream will be offered to facilitate the procedure according to individual preferences. In the control group all participants will be asked to avoid any breast stimulation during the study period.
  Arms: Intervention group

SUMMARY:
Premature Rupture of Membranes (PROM) is defined as the rupture of membranes before the onset of regular uterine contractions.

PROM occurs in approximately 10% of all pregnancies (ranging from 2.7% to 17%), with 60% to 80% of cases occurring at term. Approximately 90% of patients' experience PROM enter spontaneous labor within 24 hours, but disagreement exists among health care providers on the optimal management of women with PROM, particularly the need for and timing of inductions.

Nipple stimulation is a non-medical natural method for induction of labor. Previous studies demonstrated its effectiveness for initiating labor within 72 hours in women with favorable cervices. The actual mechanism by which such a technique results in cervical ripening is not well understood.

In this study, we aim to assess the effectiveness of nipple stimulation in gravid women with term PROM choosing expectant management.

DETAILED DESCRIPTION:
The participants in the study will be randomized into two groups of expectant management (patients desire an active approach will be excluded).

All eligible participants will be randomly allocated to either intervention or control group. They will be followed from the time of presentation with rupture of membranes at the ER and until the time of delivery. Prophylactic antibiotics will be administered after 18 hours from rupture of membranes as per departmental policy.

On admission, and after validating inclusion criteria, women will be offered to join the study. For the intervention group women will be instructed to gently massage alternate breasts, especially around the nipples for 15 minutes every 6 hours until the appearance of regular contractions but not more than 24 hours. Moist cloth or lubricating or moisturizing cream will be offered to facilitate the procedure according to individual preferences. In the control group all participants will be asked to avoid any breast stimulation during the study period.

For both groups maternal surveillance will include obstetrician assessment every 6 hours or per maternal request if painful contractions. Every assessment will include documenting maternal vital signs, sense of contraction, fetal cardiotocographic assessment and vaginal examination if painful contractions. After delivery,all participants will be requested to fill a satisfaction questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Primagravidas at term (>37) weeks having PROM
* Singleton pregnancies
* Cephalic presentation
* Unfavorable cervix (Bishop score <7)
* Desire an expectant management

Exclusion Criteria:

* Prior cesarean section/ uterine rupture / transmural uterine incision
* Non reassuring fetal heart rate monitoring (Category III)
* Signs of fetal or maternal infection
* Time elapsed since PROM > 6 hours
* Meconium or blood-stained amniotic fluid
* Any contraindication for vaginal birth

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | One year

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai Hallak, M.D, Principal Investigator — Department of Obstetrics & Gynecology, Hillel Yaffe Medical Center, Hadera; Rinat Gabbay, M.D, Study Director — Department of Obstetrics & Gynecology, Hillel Yaffe Medical Center, Hadera
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hannah ME, Ohlsson A, Farine D, Hewson SA, Hodnett ED, Myhr TL, Wang EE, Weston JA, Willan AR. Induction of labor compared with expectant management for prelabor rupture of the membranes at term. TERMPROM Study Group. N Engl J Med. 1996 Apr 18;334(16):1005-10. doi: 10.1056/NEJM199604183341601. PMID 8598837
- [Result] Cahill AG, Tuuli MG. Labor in 2013: the new frontier. Am J Obstet Gynecol. 2013 Dec;209(6):531-4. doi: 10.1016/j.ajog.2013.04.016. Epub 2013 Apr 10. PMID 23583208
- [Result] Christensson K, Nilsson BA, Stock S, Matthiesen AS, Uvnas-Moberg K. Effect of nipple stimulation on uterine activity and on plasma levels of oxytocin in full term, healthy, pregnant women. Acta Obstet Gynecol Scand. 1989;68(3):205-10. doi: 10.3109/00016348909020990. PMID 2618602
- [Result] Elliott JP, Flaherty JF. The use of breast stimulation to ripen the cervix in term pregnancies. Am J Obstet Gynecol. 1983 Mar 1;145(5):553-6. doi: 10.1016/0002-9378(83)91194-8. PMID 6338721
- [Result] Elliott JP, Flaherty JF. The use of breast stimulation to prevent postdate pregnancy. Am J Obstet Gynecol. 1984 Jul 15;149(6):628-32. doi: 10.1016/0002-9378(84)90247-3. PMID 6377899
- [Result] Hill WC, Moenning RK, Katz M, Kitzmiller JL. Characteristics of uterine activity during the breast stimulation stress test. Obstet Gynecol. 1984 Oct;64(4):489-92. PMID 6483296
- [Result] Johnson JW, Daikoku NH, Niebyl JR, Johnson TR Jr, Khouzami VA, Witter FR. Premature rupture of the membranes and prolonged latency. Obstet Gynecol. 1981 May;57(5):547-56. PMID 7219903
- [Result] Kavanagh J, Kelly AJ, Thomas J. Breast stimulation for cervical ripening and induction of labour. Cochrane Database Syst Rev. 2005 Jul 20;2005(3):CD003392. doi: 10.1002/14651858.CD003392.pub2. PMID 16034897
- [Result] Leake RD, Buster JE, Fisher DA. The oxytocin secretory response to breast stimulation in women during the menstrual cycle. Am J Obstet Gynecol. 1984 Feb 15;148(4):457-60. doi: 10.1016/0002-9378(84)90726-9. PMID 6696003
- [Result] Mishanina E, Rogozinska E, Thatthi T, Uddin-Khan R, Khan KS, Meads C. Use of labour induction and risk of cesarean delivery: a systematic review and meta-analysis. CMAJ. 2014 Jun 10;186(9):665-73. doi: 10.1503/cmaj.130925. Epub 2014 Apr 28. PMID 24778358
- [Result] Salmon YM, Kee WH, Tan SL, Jen SW. Cervical ripening by breast stimulation. Obstet Gynecol. 1986 Jan;67(1):21-4. PMID 3940333
- [Result] Viegas OA, Arulkumaran S, Gibb DM, Ratnam SS. Nipple stimulation in late pregnancy causing uterine hyperstimulation and profound fetal bradycardia. Br J Obstet Gynaecol. 1984 Apr;91(4):364-6. doi: 10.1111/j.1471-0528.1984.tb05924.x. PMID 6712896